CLINICAL TRIAL: NCT01261819
Title: "Laparoscopic" Cystoscopy Versus Traditional Cystoscopy in Patients Undergoing Minimally Invasive Hysterectomy: A Prospective Comparison Study
Brief Title: "Laparoscopic" Cystoscopy Versus Traditional Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FH Project #2142-4860
Record Dates: First submitted 2010-10-28; First posted 2010-12-17 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Lower Urinary Tract Injury
Keywords: cystoscopy, minimally invasive hysterectomy
MeSH Terms: interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- transurethral laparoscope (Experimental): These patients had cystoscopy performed with the transurethral laparoscope.
  Interventions: Device: cystoscopy
- Traditional cystoscopy (Active Comparator): These patients had cystoscopy performed with the traditional cystoscope, which is considered to be the "gold standard."
  Interventions: Device: cystoscopy

INTERVENTIONS:
Device: cystoscopy

SUMMARY:
The study aimed to compare the use of a transurethral laparoscope to the use of a traditional cystoscope for evaluation of the bladder and ureters at the time of laparoscopic hysterectomy. The hypothesis was that visual inspection of the bladder and ureters can be done safely using a transurethral laparoscope, takes less time than traditional cystoscopy, and is more cost effective than traditional cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. any female patient scheduled for a laparoscopic supracervical hysterectomy (LSH) or total laparoscopic hysterectomy (TLH) with or without adnexectomy for benign disease
2. able to comprehend and sign the informed consent form
3. able to provide clean-catch urine specimens
4. able to complete a urinary symptom questionnaire pre- and post-operatively

Exclusion Criteria:

1. participants in another research protocol involving an investigational product 30 days before planned randomization
2. pregnant women
3. patients undergoing concomitant incontinence or pelvic support procedures (e.g. transvaginal tape, transobturator tape, pelvic organ prolapse surgery)
4. patients known to have a history of recurrent urinary tract infections

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kratz, M.D., Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Winter Park and Celebration, Florida, United States

REFERENCES:
- [Derived] Kratz KG, Spytek SH, Caceres A, Lukman R, McCarus SD. A randomized, single-blinded pilot study evaluating use of a laparoscope or a cystoscope for cystoscopy during gynecologic surgery. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):606-14. doi: 10.1016/j.jmig.2012.06.002. Epub 2012 Jul 17. PMID 22818539
- See also: Publication of study — https://pubmed.ncbi.nlm.nih.gov/22818539/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transurethral Laparoscope | Traditional Cystoscopy
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transurethral Laparoscope: These patients had cystoscopy performed with the transurethral laparoscope.
  cystoscopy
- Traditional Cystoscopy: These patients had cystoscopy performed with the traditional cystoscope, which is considered to be the "gold standard."
  cystoscopy
- Total: Total of all reporting groups
Arm/Group | Transurethral Laparoscope | Traditional Cystoscopy | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (6.33) | 44.5 (5.10) | 45 (5.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 33 | 66
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (6.65) | 27.1 (5.14) | 27.85 (5.90)
Smoker (%) [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time Required to Perform Procedure (in Seconds)
Description: Time required to perform cystoscopy with a laparoscope or a cystoscope after laparoscopic hysterectomy.
Time Frame: During Procedure (Up to 15 minutes)
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Transurethral Laparoscope | Traditional Cystoscopy
Number analyzed (Participants) | 33 | 33
seconds | 137 [21.1 to 249.9] | 451 [204.63 to 697.37]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study January-July 2009, and up to 6 weeks after the surgical intervention for each subject.
Arm/Group | Transurethral Laparoscope | Traditional Cystoscopy
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 1/33 | 6/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transurethral Laparoscope (N=33) | Traditional Cystoscopy (N=33)
bladder discomfort/pain (Renal and urinary disorders) | 0 | 2
hematoma (Renal and urinary disorders) | 0 | 1
Postoperative Urinary Tract Infection (UTI) (Renal and urinary disorders) | 0 | 2
Vaginal bleed (Reproductive system and breast disorders) | 0 | 1
Trocar-site bleed (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes